CLINICAL TRIAL: NCT04548284
Title: Periorbitally Injected Glucocorticoids for Mild TAO: A Randomized Controlled Study
Brief Title: Study of Therapeutic Value of Periorbital Injection of Glucocorticoid in Mild TAO
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Huasheng Yang, Principal Investigator, Clinical Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: yanghs202009
Record Dates: First submitted 2020-09-07; First posted 2020-09-14 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Thyroid Associated Ophthalmopathy
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — Glucocorticoids

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Periorbitally Injected Glucocorticoids (Experimental): Glucocorticoids periorbital injection. Once every 3 weeks, the number of injections was determined according to the condition of the eyes during the follow-up.
  Interventions: Drug: Glucocorticoids
- Observe (No Intervention): Observe and wait.

INTERVENTIONS:
Drug: Glucocorticoids — Periorbital injection of glucocorticoid. Once every 3 weeks, the number of injections was determined according to the condition of the eyes during the follow-up.
  Arms: Periorbitally Injected Glucocorticoids

SUMMARY:
The purpose of this study is to determine whether periorbital injection of glucocorticoid is effective and necessary in the treatment of mild TAO.

ELIGIBILITY:
Inclusion Criteria:

General conditions:

1. clinically diagnosed as thyroid disease;
2. able and willing to participate in clinical trials and ensure regular follow-up.

Eye condition:

1. patients with monocular disease diagnosed by TAO;
2. EUGOGO/NOSPECS grade was mild and CAS score was less than 3;
3. the course of eye disease was less than 12mo and had not been treated in the past.

Exclusion Criteria:

General situation:

1. patients with poor blood glucose control in recent 3 months, glycosylation ≥ 10% ;
2. blood pressure still fluctuated > 180/110mmHg after medication;
3. obvious liver and kidney insufficiency;
4. contraindications for the use of glucocorticoids (peptic ulcer, osteoporosis, severe infection, psychosis, etc.);
5. patients with severe abnormal blood coagulation;
6. patients with other systemic immune diseases;
7. any uncontrollable clinical problems (severe mental, neurological, cardiovascular, respiratory and other systemic diseases and malignant tumors);
8. history of chronic infection;
9. pregnant and lactating women.

Eye conditions:

1. B-ultrasound or CT, MRI found other diseases causing exophthalmos (intraorbital space occupying lesion, inflammatory pseudotumor, neurofibroma, etc.);
2. moderate to severe TAO, in either eye requiring local or systemic treatment;
3. periorbital infectious diseases, hemorrhagic diseases;
4. uveitis, glaucoma, high myopia, diabetic retinopathy and other eye diseases.
5. those who studied the eyes who had a history of arbitrary surgery;
6. those who were considered by the researchers to be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change of Clinical Activity Score (CAS) score | baseline、3months、6months、9months、12months
  Comparison of CAS scores before and after treatment in each arm and an inter-arm. The range of CAS scores is 0-7, with 3 as the boundary. The higher the score, the higher the activity.
Change of NOSPECS score | baseline、3months、6months、9months、12months
  Comparison of NOSPECS scores before and after treatment in each arm and an inter-arm. The NOSPECS score was 0-6. The higher the score, the higher the severity.

SECONDARY OUTCOMES:
adverse events | baseline、3months、6months、9months、12months
  Comparison of adverse events rate in each arm and an inter-arm.
Quality of life questionnaires (GO-QoL) | baseline、3months、6months、9months、12months
  Comparison of Graves' ophthalmopathy Quality of life questionnaire (GO-QOL) scores before and after treatment in each arm and an inter-arm. The GO-QOL score is between 0 and 100. The higher the score, the better the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Huasheng Yang, Doctor, Study Chair — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided